CLINICAL TRIAL: NCT05936476
Title: Influence of Different Types of Maxillomandibular Deformities on the Nutritional Status of Individuals: A Cross-sectional Study
Brief Title: Impact of Maxillomandibular Deformities on Individuals' Nutritional Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist Prof., Marmara University
Other Study IDs: MUDHF_ORT_SBF_01
Record Dates: First submitted 2023-06-23; First posted 2023-07-07 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Maxillofacial Abnormalities
Keywords: Orthognathic surgery; Nutritional status; Angles classification
MeSH Terms: conditions — Maxillofacial Abnormalities; Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Skeletal Class I (Control Group)
- Skeletal Class II: Class II malocclusion is characterized by the upper jaw (maxilla) being positioned more forward in relation to the lower jaw (mandible), resulting in an overbite.
- Skeletal Class III: Class III malocclusion is characterized by the lower jaw (mandible) being positioned more forward in relation to the upper jaw (maxilla), resulting in an underbite.
- Anterior Open Bite: Anterior open bite is characterized by a lack of vertical overlap or contact between the upper and lower front teeth when the back teeth are in contact (occlusion).

SUMMARY:
This cross-sectional study explores the influence of various types of maxillomandibular deformities on the nutritional status of individuals. Maxillomandibular deformities, which involve the misalignment of the upper and lower jaws, can significantly affect oral functionality, potentially leading to nutritional deficiencies due to compromised food intake. By analyzing the dietary habits and nutritional health of a diverse group of individuals with these deformities, the study seeks to establish the correlation between the severity of the deformity and the individual's nutritional status. Findings from this research can provide a deeper understanding of the additional health risks that maxillomandibular deformities pose and help in the development of nutritional guidelines specifically tailored for individuals suffering from these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 45 years old
* Individuals who are not currently undergoing orthodontic treatment and have a complete set of teeth, excluding wisdom teeth.
* Citizens of the Republic of Turkey
* Able to read and write in Turkish language
* Able to understand and follow the questionnaire instructions
* Willing to participate in the study

Exclusion Criteria:

* Individuals above 45 years old
* Unwilling to sign the informed consent for participation in the study
* Unwilling to answer all the questionnaire items
* Individuals with a chronic disease that requires a specific diet
* Individuals with any eating disorders
* Pregnant and/or nursing individuals
* Individuals with cognitive impairment to a degree that would prevent giving clear and accurate responses will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include adult individuals aged 18 to 45 years who are citizens of the Republic of Turkey. At the time of enrollment, these individuals should not be undergoing any orthodontic treatment and should have a complete set of teeth, excluding wisdom teeth. They should possess basic reading and writing skills in the Turkish language and be able to comprehend and comply with the instructions for completing the questionnaire. Additionally, their voluntary participation in the study will be required.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Dietary Intake Record (24-hour recall method) | Day 1
  This measure involves recalling all the food and beverages consumed by an individual over the previous day. The 24-hour recall will be conducted through detailed questions asked by the researchers of the study to obtain more precise information about the individual's consumption. The collected dietary intake records will be analyzed using the Computer-Assisted Nutrition Program, Nutrition Information Systems Package Program (BEBIS). The quantities of nutrients included in the meals will be calculated using the "Standard Meal Recipes" book, and serving sizes will be determined using the "Food and Meal Photo Catalog" book.
Assessment of Diet Quality using Healthy Eating Index (HEI-2015) | Day 1
  The Healthy Eating Index (HEI) is a tool developed by the USDA's Center for Nutrition Policy and Promotion to assess the quality of an individual's diet. The HEI-2015, the most recent version, consists of 13 components that evaluate both adequacy and moderation of dietary intake. Nine components focus on the consumption of essential nutrients and food groups, including fruits, vegetables, whole grains, dairy, protein foods, and fatty acids. The remaining four components assess the intake of less healthy items, such as refined grains, added sugars, sodium, and saturated fats. Each component is assigned a score, and the total score can range from 0 to 100. Higher scores indicate better adherence to recommended dietary guidelines. The HEI-2015 score is classified into three categories: scores below 50 indicate poor diet quality, scores between 51 and 80 suggest a need for dietary improvements, and scores above 80 indicate good diet quality.

SECONDARY OUTCOMES:
Antropometric measurements - Height | Day 1
  Height will be measured with the participant standing barefoot and upright, with the head, back, and hips touching the wall. Height will be measured with a meter and recorded in centimeters. The measurement will be taken using a wall-mounted stadiometer.
Body Composition | Day 1
  Body composition analysis will be performed with the Tanita DC-360 device that performs bioelectrical impedance analysis (BIA). The analysis report includes body weight (kg), body water mass (kg), body fat mass (kg) and body muscle mass (kg). This method is non-invasive and provides body composition data in less than 1 minute of measurement.
Waist Circumference Measurement | Day 1
  Waist circumference measurement will be taken from the thinnest point of the participant, below the ribs and above the belly. During the measurement, the individual will be standing and exhaling in a relaxed state. The measurement tape will be placed around the waist in a horizontal line and will be measured in cm.
Body Mass Index Measurement | Day 1
  The Body Mass Index will be calculated as weight (kg)/height (m2). The WHO classification will be used to categorize: · BMI < 18.5: Underweight · BMI 18.5 - 24.9: Normal · BMI 25.0 - 29.9: Overweight · BMI 30.0 - 34.9: Class I Obesity · BMI 35.0 - 39.
Physical Activity Level | Day 1
  The physical activity levels of the individuals included in the study will be evaluated using the short form of the International Physical Activity Questionnaire (IPAQ). The short form of the International Physical Activity Questionnaire (7 questions) is used to evaluate physical activity in 4 areas including leisure time, household, work, and transportation over a seven-day period. Physical activity level is classified as active, moderately active, and inactive based on general scores. The IPAQ short form, developed with the support of the World Health Organization (WHO) and the US Centers for Disease Control and Prevention (CDC), has had its validity and reliability study performed in Turkey by Sağlam et al. It provides information about the time individuals spend in light, moderate, and intense activities, as well as sitting duration.
Chewing Ability Assessment | Day 1
  Chewing ability can be evaluated both objectively and subjectively. Subjective evaluation includes assessment using questionnaires and scales, and it is stated that questionnaires are the most effective tools in evaluating chewing ability in complete denture patients. In this study, a questionnaire form consisting of open-ended and closed-ended questions will be used to determine individuals' chewing difficulties. Open-ended questions will inquire about foods that are difficult to chew and the methods used to consume these foods. In follow-up interviews, closed-ended questions about the ability to chew foods previously listed will be asked as "easy to chew", "experiencing some difficulty", "experiencing great difficulty/cannot chew at all". If the individual says "I have a little or a lot of difficulty" in at least two of the hard foods and "a little or a lot of difficulty" in at least four of the soft foods, it will be evaluated as "there is difficulty in chewing".

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2017 Diet Collaborators. Health effects of dietary risks in 195 countries, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 May 11;393(10184):1958-1972. doi: 10.1016/S0140-6736(19)30041-8. Epub 2019 Apr 4. PMID 30954305
- [Background] Micha R, Penalvo JL, Cudhea F, Imamura F, Rehm CD, Mozaffarian D. Association Between Dietary Factors and Mortality From Heart Disease, Stroke, and Type 2 Diabetes in the United States. JAMA. 2017 Mar 7;317(9):912-924. doi: 10.1001/jama.2017.0947. PMID 28267855
- [Background] Backholer K, Spencer E, Gearon E, Magliano DJ, McNaughton SA, Shaw JE, Peeters A. The association between socio-economic position and diet quality in Australian adults. Public Health Nutr. 2016 Feb;19(3):477-85. doi: 10.1017/S1368980015001470. Epub 2015 May 20. PMID 25989940
- [Background] Reedy J, Krebs-Smith SM, Miller PE, Liese AD, Kahle LL, Park Y, Subar AF. Higher diet quality is associated with decreased risk of all-cause, cardiovascular disease, and cancer mortality among older adults. J Nutr. 2014 Jun;144(6):881-9. doi: 10.3945/jn.113.189407. Epub 2014 Feb 26. PMID 24572039
- [Background] de Andrade SC, de Azevedo Barros MB, Carandina L, Goldbaum M, Cesar CL, Fisberg RM. Dietary quality index and associated factors among adolescents of the state of Sao Paulo, Brazil. J Pediatr. 2010 Mar;156(3):456-60. doi: 10.1016/j.jpeds.2009.09.066. Epub 2009 Dec 14. PMID 20004911
- [Background] Moynihan P, Thomason M, Walls A, Gray-Donald K, Morais JA, Ghanem H, Wollin S, Ellis J, Steele J, Lund J, Feine J. Researching the impact of oral health on diet and nutritional status: methodological issues. J Dent. 2009 Apr;37(4):237-49. doi: 10.1016/j.jdent.2008.12.003. Epub 2009 Jan 20. PMID 19157673
- [Background] Koksal E, Karacil Ermumcu MS, Mortas H. Description of the healthy eating indices-based diet quality in Turkish adults: a cross-sectional study. Environ Health Prev Med. 2017 Mar 20;22(1):12. doi: 10.1186/s12199-017-0613-z. PMID 29165107